CLINICAL TRIAL: NCT05512819
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE GIVEN IN A SERIES OF 3 INFANT DOSES AND 1 TODDLER DOSE IN INFANTS IN INDIA AND TAIWAN
Brief Title: A Study to Describe the Safety and Immunogenicity of 20vPnC in Infants in India and Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B7471024; NCT05512819 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20-valent pneumococcal conjugate vaccine (Experimental): Pneumococcal conjugate vaccine (20vPnC)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine
- 13-valent pneumococcal conjugate vaccine (Active Comparator): Pneumococcal conjugate vaccine (13vPnC)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — 20-valent pneumococcal conjugate vaccine
  Arms: 20-valent pneumococcal conjugate vaccine
Biological: 13-valent pneumococcal conjugate vaccine — 13-valent pneumococcal conjugate vaccine
  Arms: 13-valent pneumococcal conjugate vaccine

SUMMARY:
The purpose of this study is to understand the safety and effects of a study vaccine (20vPnC) in infants and toddlers.

This study is enrolling participants who are:

* Born after at least 36 weeks of pregnancy and about 2 months of age at the time of entering the study
* Have a bodyweight of at least 3 kg

Participants will receive either the study vaccine (20vPnC) or a licensed vaccine (13vPnC) as a 4-dose schedule as a shot in the muscle. Participants will receive Dose 1 on study day 1. Dose 2 will be given 28-70 days after Dose 1, and Dose 3 will be given 28-70 days after Dose 2. Dose 4 will be given at 365-455 days (approximately 12-15 months) of age.

Participation in the study will take approximately 15 months, during which participants will come to the study clinic for 6 times. The study team will ask questions about the participant's health and take some blood samples during the visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born at ≥36 weeks of gestation and approximately 2 months of age at the time of consent
* Healthy infants determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study
* Weight of 3.0 kg or greater at the time of randomization

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of 13vPnC, 20vPnC, or any other diphtheria toxoid-containing vaccine.
* Major known congenital malformation or serious chronic disorder
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study intervention administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study
* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.

Ages: 42 Days to 84 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 541 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in India and Taiwan with local reactions (redness, swelling, and pain at the injection site), separately by country | Day 7
  Prompted local reactions after each dose
Percentage of participants in India and Taiwan with systemic events (fever, decreased appetite, drowsiness/increased sleep, and irritability), separately by country | Day 7
  Prompted systemic reactions after each dose
Percentage of participants in India and Taiwan with adverse events (AEs) from Dose 1 through 1 month after Dose 3 in each group, separately by country | Dose 1 to 1 month after Dose 3
  Adverse events occurring from Dose 1 to 1 month after Dose 3 in each group
Percentage of participants from India and Taiwan with AEs from Dose 4 through 1 month after Dose 4 in each group, separately by country | Dose 4 to 1 month after Dose 4
  Adverse events occurring from Dose 4 to 1 month after Dose 4 in each group
Percentage of participants in India and Taiwan with SAEs from Dose 1 through 1 month after Dose 4 in each group, separately by country | Dose 1 to 1 month after Dose 4
  SAEs occurring up to 1 month after Dose 4 in each group
GMCs of serotype-specific IgG concentrations in Indian participants 1 month after Dose 4 in each vaccine group | 1 month after Dose 4
  IgG GMCs for the 20vPnC serotypes 1 month after Dose 4, Indian participants only

SECONDARY OUTCOMES:
Geometric mean concentrations (GMCs) of serotype-specific IgG concentrations 1 month after Dose 3 in each vaccine group, separately by country | 1 month after Dose 3
  IgG GMCs for the 20vPnC serotypes 1 month after Dose 3
Percentages of participants in India and Taiwan with predefined serotype-specific IgG concentration for the 20vPnC serotypes at approximately 1 month after Dose 3 in each vaccine group, separately by country | 1 month after Dose 3
  IgG concentrations for 20vPnC serotypes 1 month after Dose 3
GMCs of serotype-specific IgG concentrations in Taiwanese participants 1 month after Dose 4 in each vaccine group | 1 month after Dose 4
  IgG GMCs for the 20vPnC serotypes 1 month after Dose 4, Taiwanese participants only
Percentages of participants in India and Taiwan with predefined serotype-specific IgG concentrations for the 20vPnC serotypes at approximately 1 month after Dose 4 in each vaccine group, separately by country | 1 month after Dose 4
  IgG concentrations for 20vPnC serotypes 1 month after Dose 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- India (6):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - BGS Global Institute of Medical Sciences (BGSGIMS), Bangalore, Karnataka
  - Bharati Vidyapeeth {Deemed to be University) Medical College Hospital & Research Centre, Pune, Maharashtra
  - Maulana Azad Medical College and Associated with Lok Nayak Hospital, New Delhi, National Capital Territory of Delhi
  - Jawahar Lal Nehru Medical College, Ajmer, Rajasthan
  - Institute of Child Health, Kolkata, West Bengal
- Taiwan (5):
  - Hsinchu Mackay Memorial Hospital, Hsinchu, Hsinchu
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471024